CLINICAL TRIAL: NCT04490317
Title: CARbon monoxidE intoxiCatiOn in Korea: Prospective Cohort (CARE CO Cohort)
Status: Recruiting | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Yong Sung Cha, Assistant Professor, Wonju Severance Christian Hospital
Other Study IDs: CARE CO cohort
Record Dates: First submitted 2020-07-21; First posted 2020-07-29 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Carbon Monoxide Poisoning; Myocardial Injury; Neurologic Deficits; Image, Body; Therapy; Prognostic Factors; Complications
MeSH Terms: conditions — Carbon Monoxide Poisoning; Neurologic Manifestations | interventions — Echocardiography; Clinical Laboratory Techniques; Hyperbaric Oxygenation; Hypothermia, Induced

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute CO poisoning: A diagnosis of CO poisoning is made according to medical history and carboxyhemoglobin >5% (>10% in smokers).
  Interventions: Diagnostic Test: Cardiac MRI; Procedure: Hyperbaric oxygen therapy

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — 1. Cardiac MRI be taken to CO poisoned patients
  2. Cardiac CT be taken to CO poisoned patients
  3. TTE be taken to CO poisoned patients
  4. Brain MRI be taken to CO poisoned patients
  5. Neurocognitive function tests be taken to CO poisoned patients
  6. Laboratory tests be taken to CO poisoned patients
  Other Names: Cardiac CT; Transthoracic echocardiography (TTE); Brain MRI; Neurocognitive function tests; Laboratory tests
Procedure: Hyperbaric oxygen therapy — 1. Hyperbaric oxygen therapy be used for CO poisoned patients
  2. Therapeutic hypothermia be used for CO poisoned patients
  Other Names: Therapeutic hypothermia

SUMMARY:
This prospective cohort study enrolls subjects who experience carbon monoxide (CO) poisoning. The purpose of the study is to evaluate therapeutic effects of various treatments and short and long-term outcomes in CO poisoned patients. In addition, complications of brain and heart susceptible to CO are investigated through various ways and the association between complications and the patient's prognosis is also investigated. All subjects will be regularly monitored by physicians participating in this study.

DETAILED DESCRIPTION:
This prospective cohort study enrolls subjects who experience CO poisoning. The purpose of the study is to evaluate therapeutic effects of various treatments, including hyperbaric oxygen therapy (HBO), therapeutic hypothermia (TH), and additional drugs, and short and long-term outcomes, such as neurocognitive sequelae or mortality, in CO poisoned patients. In addition, complications of brain and heart susceptible to CO are investigated through a variety of ways, such as magnetic resonance image (MRI), computed tomography (CT), ultrasound, and laboratory test, and the association between various complications and the patient's prognosis is also investigated. All subjects will be regularly monitored by physicians participating in this study.

ELIGIBILITY:
Inclusion Criteria:

* Acute CO poisoning

Exclusion Criteria:

* Declined to enrollment in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Acute CO poisoning
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-07-29 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Therapeutic response to HBO at 1 month | At 1 month after CO exposure
  Therapeutic response to HBO according to times from rescue to first HBO and frequency and pressure of HBO at 1 month after CO exposure
Therapeutic response to HBO at 6 months | At 6 months after CO exposure
  Therapeutic response to HBO according to times from rescue to first HBO and frequency and pressure of HBO at 6 months after CO exposure
Predictors and model development for participants with poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure evaluated by such as neurocognitive function tests | Within 1 month after CO exposure
  Predictors and model development for poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure evaluated by tools, such as global deterioration scale (GDS) or Carbon Monoxide Neuropsychological Screening Battery (CONSB), etc, through variables, such as clinical features, laboratory tests, or imaging study that can be investigated within 1 month
Predictors and model development for participants with poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure evaluated by such as neurocognitive function tests | Within 1 month after CO exposure
  Predictors and model development for poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure evaluated by tools, such as global deterioration scale (GDS) or Carbon Monoxide Neuropsychological Screening Battery (CONSB), etc, through variables, such as clinical features, laboratory tests, or imaging study that can be investigated within 1 month
Predictors and model development for participants with poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure evaluated by such as neurocognitive function tests | Within 1 month after CO exposure
  Predictors and model development for poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure evaluated by tools, such as global deterioration scale (GDS) or Carbon Monoxide Neuropsychological Screening Battery (CONSB), etc, through variables, such as clinical features, laboratory tests, or imaging study that can be investigated within 1 month

SECONDARY OUTCOMES:
Therapeutic response to HBO at 12 months | At 12 months after CO exposure
  Therapeutic response to HBO according to times from rescue to first HBO and frequency and pressure of HBO at 12 months after CO exposure
Therapeutic response to TH combined with HBO at 1 month | At 1 month after CO exposure
  Therapeutic response to TH combined with HBO in acute severe CO poisoning at 1 month after CO exposure
Therapeutic response to TH combined with HBO at 6 months | At 6 months after CO exposure
  Therapeutic response to TH combined with HBO in acute severe CO poisoning at 6 months after CO exposure
Therapeutic response to TH combined with HBO at 12 months | At 12 months after CO exposure
  Therapeutic response to TH combined with HBO in acute severe CO poisoning at 12 months after CO exposure
Therapeutic response to HBO according to presence of apolipoprotein E4 at 1 month | At 1 month after CO exposure
  Therapeutic response to HBO according to presence of apolipoprotein E4 genotype at 1 month after CO exposure
Therapeutic response to HBO according to presence of apolipoprotein E4 at 6 months | At 6 months after CO exposure
  Therapeutic response to HBO according to presence of apolipoprotein E4 genotype at 6 months after CO exposure
Therapeutic response to HBO according to presence of apolipoprotein E4 at 12 months after CO exposure | At 12 months after CO exposure
  Therapeutic response to HBO according to presence of apolipoprotein E4 genotype at 12 months after CO exposure
Cardiac injury evaluated by cardiac MRI in acute phase | Within 1 month after CO exposure
  Cardiac injury related to CO poisoning evaluated by cardiac MRI in acute phase
Cardiac injury evaluated by cardiac MRI in chronic phase | Follow-up cardiac MRI (at 4-8 months after CO exposure)
  Cardiac injury related to CO poisoning evaluated by cardiac MRI in chronic phase
Cardiac injury evaluated by cardiac CT | Within 1 month after CO exposure
  Cardiac injury evaluated by cardiac CT in CO poisoning
Cardiac injury evaluated by TTE in acute phase | Within 14 days after CO exposure
  Cardiac injury related to CO poisoning evaluated by TTE in acute phase
Cardiac injury evaluated by TTE in chronic phase | Within 4-8 months after CO exposure
  Cardiac injury related to CO poisoning evaluated by TTE in chronic phase
Brain injury evaluated by brain imaging modality related to CO poisoning | Within 6 months after CO exposure
  Brain injury evaluated by brain MRI in CO poisoning
Brain injury related to CO poisoning | Within 6 months after CO exposure
  Brain injury evaluated by laboratory tests in CO poisoning
Association between presence of cardiac injury, which is evaluated by cardiac enzyme or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure | Outcomes at 1 month after CO exposure
  Association between presence of cardiac injury, which is evaluated by electrocardiogram, cardiac enzyme, or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure
Association between presence of cardiac injury, which is evaluated by cardiac enzyme or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure | Outcomes at 6 months after CO exposure
  Association between presence of cardiac injury, which is evaluated by electrocardiogram, cardiac enzyme, or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure
Association between presence of cardiac injury, which is evaluated by cardiac enzyme or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure | Outcomes at 12 months after CO exposure
  Association between presence of cardiac injury, which is evaluated by electrocardiogram, cardiac enzyme, or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure
Association between presence of cardiac injury, which is evaluated by cardiac enzyme or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 5 years after CO exposure | Outcomes at 5 years after CO exposure
  Association between presence of cardiac injury, which is evaluated by electrocardiogram, cardiac enzyme, or cardiac imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 5 years after CO exposure
Association between presence of brain injury, which is evaluated by brain imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure evaluated by neurocognitive function tests | Outcomes at 1 month after CO exposure
  Association between presence of brain injury, which is evaluated by brain MRI, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure evaluated by such as GDS or CONSB, etc
Association between presence of brain injury, which is evaluated by brain imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure evaluated by neurocognitive function tests | Outcomes at 6 months after CO exposure
  Association between presence of brain injury, which is evaluated by brain MRI, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure evaluated by such as GDS or CONSB, etc
Association between presence of brain injury, which is evaluated by brain imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure evaluated by neurocognitive function tests | Outcomes at 12 months after CO exposure
  Association between presence of brain injury, which is evaluated by brain MRI, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure evaluated by such as GDS or CONSB, etc
Association between presence of brain injury, which is evaluated by brain imaging studies, and poor outcome including mortality, and neurocognitive and psychological sequelae at 5 years after CO exposure evaluated by neurocognitive function tests | Outcomes at 5 years after CO exposure
  Association between presence of brain injury, which is evaluated by brain MRI, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 5 years after CO exposure evaluated by such as GDS or CONSB, etc
Association between presence of brain injury, which is evaluated by laboratory tests, and poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure evaluated by neurocognitive function tests | Outcomes at 1 month after CO exposure
  Association between presence of brain injury, which is evaluated by laboratory tests, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 1 month after CO exposure evaluated by such as GDS or CONSB, etc
Association between presence of brain injury, which is evaluated by laboratory tests, and poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure evaluated by neurocognitive function tests | Outcomes at 6 months after CO exposure
  Association between presence of brain injury, which is evaluated by laboratory tests, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 6 months after CO exposure evaluated by such as GDS or CONSB, etc
Association between presence of brain injury, which is evaluated by laboratory tests, and poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure evaluated by neurocognitive function tests | Outcomes at 12 months after CO exposure
  Association between presence of brain injury, which is evaluated by laboratory tests, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 12 months after CO exposure evaluated by such as GDS or CONSB, etc
Association between presence of brain injury, which is evaluated by laboratory tests, and poor outcome including mortality, and neurocognitive and psychological sequelae at 5 years after CO exposure evaluated by neurocognitive function tests | Outcomes at 5 years after CO exposure
  Association between presence of brain injury, which is evaluated by laboratory tests, etc, and poor outcome including mortality, and neurocognitive and psychological sequelae at 5 years after CO exposure evaluated by such as GDS or CONSB, etc
Therapeutic response to drugs at 1 month | At 1 month after CO exposure
  Therapeutic response to additional drug including steroid at 1 month after CO exposure
Therapeutic response to drugs at 6 months | At 6 months after CO exposure
  Therapeutic response to additional drug including steroid at 6 months after CO exposure
Therapeutic response to drugs at 12 months | At 12 months after CO exposure
  Therapeutic response to additional drug including steroid at 12 months after CO exposure
Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae after CO poisoning at 1 month | At 1 month after CO exposure
  Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae evaluated by, such as GDS or CONSB, etc, after CO poisoning at 1 month after CO exposure
Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae after CO poisoning at 6 months | At 6 months after CO exposure
  Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae evaluated by, such as GDS or CONSB, etc, after CO poisoning at 6 months after CO exposure
Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae after CO poisoning at 12 months | At 12 months after CO exposure
  Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae evaluated by, such as GDS or CONSB, etc, after CO poisoning at 12 months after CO exposure
Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae after CO poisoning at 5 years | At 5 years after CO exposure
  Prevalence of poor outcomes including mortality, and neurocognitive and psychological sequelae evaluated by, such as GDS or CONSB, etc, after CO poisoning at 5 years after CO exposure
Organ injury related to CO poisoning | Within 6 months after CO exposure
  Organ injury, such as lung, kidney, liver, pancreas, or bowel, etc, related to CO poisoning
Complications related to CO poisoning | Within 6 months after CO exposure
  Complications, such as pulmonary thromboembolism or rhabdomyolysis, etc, related to CO poisoning
Effect of HBO for delayed neurocognitive and psychological dysfunction at 1 year after onset | Within 1 year after delayed neurocognitive and psychological sequelae onset
  Effect of HBO for patient with delayed neurocognitive and psychological sequelae at 1 year after sequelae onset
Effect of HBO for delayed neurocognitive and psychological dysfunction at 2 years after onset | Within 2 years after delayed neurocognitive and psychological sequelae onset
  Effect of HBO for patient with delayed neurocognitive and psychological sequelae at 2 years after sequelae onset
Validation of methods evaluating neurocognitive and psychological outcomes | Within 6 months after CO exposure
  Validation of methods evaluating neurocognitive and psychological outcomes within 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yong Sung Cha, MD, Principal Investigator — Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea

REFERENCES:
- [Derived] Ahn GJ, Lee S, Heo YW, Cha YS. Mortality Risks and Causes in Previous Carbon Monoxide Poisoning: A Nationwide Population-Based Cohort Study. Crit Care Med. 2024 Dec 1;52(12):1866-1876. doi: 10.1097/CCM.0000000000006414. Epub 2024 Sep 18. PMID 39298511